CLINICAL TRIAL: NCT04547140
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of Liquid Alpha1-Proteinase Inhibitor (Human) Plus Standard Medical Treatment (SMT) Versus Placebo Plus SMT in Hospitalized Subjects With COVID-19
Brief Title: Study to Evaluate the Safety and Efficacy of Liquid Alpha1-Proteinase Inhibitor (Human) in Hospitalized Participants With Coronavirus Disease (COVID-19)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Stopped for Futility
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC2006
Record Dates: First submitted 2020-09-10; First posted 2020-09-14 (Actual); Results first posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: Coronavirus Disease; Severe acute respiratory syndrome coronavirus 2; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — alpha 1-Antitrypsin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liquid Alpha1-Proteinase Inhibitor + Standard Medical Treatment (Experimental): Participants received the first intravenous (IV) infusion of liquid alpha1-proteinase inhibitor (human) 120 milligrams per kilogram (mg/kg), based on body weight on Day 1, followed by second liquid alpha1-proteinase inhibitor (human) dose of 120 mg/kg based on body weight, on Day 8 (second dose was not mandatory and was given at the principal investigator's [PI] discretion). Participants also received all standard of care interventions while hospitalized, from Day 1 to Day 29.
  Interventions: Biological: Liquid Alpha1-Proteinase Inhibitor (Human); Drug: Standard Medical Treatment
- Placebo + Standard Medical Treatment (Placebo Comparator): Participants received IV infusions of 0.9% normal saline of commensurate volume to that of liquid alpha1-proteinase inhibitor as placebo on Day 1 and Day 8 (Day 8 was not mandatory and was given at the PI's discretion). Participants also received all standard of care interventions while hospitalized, from Day 1 to Day 29.
  Interventions: Drug: Placebo; Drug: Standard Medical Treatment

INTERVENTIONS:
Biological: Liquid Alpha1-Proteinase Inhibitor (Human) — Intravenous infusion 120 mg/kg
  Other Names: Alpha1-proteinase inhibitor
  Arms: Liquid Alpha1-Proteinase Inhibitor + Standard Medical Treatment
Drug: Placebo — Intravenous infusion
  Other Names: 0.9% Normal Saline
  Arms: Placebo + Standard Medical Treatment
Drug: Standard Medical Treatment — SMT

SUMMARY:
The purpose of the study is to determine if Liquid Alpha1-Proteinase Inhibitor (Human) (Liquid Alpha1-PI) plus SMT can reduce the proportion of participants dying or requiring intensive care unit (ICU) admission on or before Day 29 or who are dependent on high flow oxygen devices or invasive mechanical ventilation on Day 29 versus placebo plus SMT in hospitalized participants with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized male or female participant ≥ 18 years of age at time of screening who is being treated for COVID-19. Participants must be screened within 48 hours (≤ 48 hours) of hospital admission.
2. Has laboratory-confirmed novel coronavirus {SARS-CoV-2} infection as determined by qualitative polymerase chain reaction (PCR) (reverse transcriptase [RT]-PCR), or other commercial or public health assay approved by regulatory authorities as a diagnostic test for COVID-19 in any specimen during the current hospital admission OR 96 hours prior to the hospital admission date and prior to randomization (the SARS-CoV-2 test results must be performed by a hospital laboratory and the documentation available).
3. COVID-19 illness (symptoms) of any duration, including both of the following: a) Radiographic infiltrates by imaging (chest X-Ray, computed tomography (CT) scan, etc.) and/or clinical assessment (evidence of rales/crackles on exam) with peripheral oxygen saturation by pulse oximetry (SpO2) <94% on room air; b) Any one of the following related to COVID-19: i. Ferritin > 400 nanogram per milliliter (ng/mL), ii. lactate dehydrogenase (LDH) > 300 units per liter (U/L), iii. D-Dimers > reference range, or iv. C-reactive protein (CRP) > 40 milligram per liter (mg/L).
4. Participant provides informed consent prior to initiation of any study procedures.
5. Female participants of childbearing potential (and males with female partners of childbearing potential) must agree to use of acceptable contraception methods during study (example, oral, injectable, or implanted hormonal methods of contraception, placement of an intrauterine device or intrauterine system, condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization, or true abstinence) throughout the study.

Exclusion Criteria:

1. Participants requiring invasive mechanical ventilation or ICU admission or with partial pressure of arterial oxygen/ fraction of inspired oxygen (PaO2/FIO2) ≤ 150 mmHg (i.e., arterial oxygen in millimeter of mercury (mmHg) divided by fraction inspired oxygen concentration [example, 0.21 for room air]).
2. Clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may place the participant at undue medical risk.
3. The participant has had a known serious anaphylactic reaction to blood, any blood-derived or plasma product, or known selective immunoglobulin A (IgA) deficiency with anti-IgA antibodies.
4. A medical condition in which the infusion of additional fluid is contraindicated (example, decompensated congestive heart failure or renal failure with fluid overload). This includes currently uncontrolled congestive heart failure New York Heart Association Class III or IV stage heart failure.
5. Shock that is unresponsive to fluid challenge and/or multiple vasopressors and accompanied by multiorgan failure considered not able to be reversed by the Principal Investigator.
6. Known alpha-1 antitrypsin deficiency for which the participant is already receiving alpha1-proteinase inhibitor augmentation therapy.
7. Women who are pregnant or breastfeeding. Female participants of child-bearing potential must have a negative test for pregnancy blood or urine human chorionic gonadotropin (HCG)-based assay at screening/baseline visit.
8. Participants for whom there is limitation of therapeutic effort such as "Do not resuscitate" status.
9. Currently participating in another interventional clinical trial with investigational medical product or device.
10. Participants previously requiring long-term oxygen therapy (home oxygen therapy).
11. History (within the last 2 years) of myocardial infarction, unstable angina, stroke or transient ischemic attacks, pulmonary embolism or deep venous thrombosis.
12. Participant has medical condition (other than COVID-19) that is projected to limit lifespan to ≤ 1 year.
13. Systolic blood pressure < 100 mm Hg or > 160 mm Hg (uncontrolled hypertension) at the time of Screening.
14. Alanine aminotransferase (ALT) ≥ 2 times the upper limit of normal (ULN).
15. Any elevation of total bilirubin at the time of Screening.
16. Estimated glomerular filtration rate (eGFR) < 45 mL/min (or participant is dependent on dialysis/renal replacement therapy) at the time of Screening. eGFR is calculated by the Cockcroft-Gault equation.
17. Hemoglobin < 10 g/dL at the time of Screening.
18. Absolute neutrophil count < 1000/mm^3 at the time of Screening.
19. Platelet count < 75,000/mm^3 at the time of Screening.
20. Participant has history of drug or alcohol abuse within the past 24 months.
21. Participant is unwilling to commit to follow-up visits.
22. Known history of prothrombin gene mutation 20210, homozygous Factor V Leiden mutations, antithrombin III deficiency, protein C deficiency, protein S deficiency or antiphospholipid syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (10):
  - Birmingham VA, Birmingham, Alabama
  - St. Joseph's Hospital, Phoenix, Arizona
  - University of Miami Hospital, Miami, Florida
  - Sparrow Hospital, Lansing, Michigan
  - Hannibal Clinic, Hannibal, Missouri
  - Kansas City VA, Kansas City, Missouri
  - CHI Health Center, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York
  - Memphis VA, Memphis, Tennessee
  - University of Utah, Salt Lake City, Utah
- Brazil (6):
  - AngioCor Blumenau, Blumenau, Santa Catarina
  - Sociedade Literaria e Caritativa Santo Agostinho, Criciúma, Santa Catarina
  - Universidade Estadual São Paulo - Campus de Botucatu, Botucatu, São Paulo
  - Hospital Dia do Pulmão, Blumenau
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo
- Chile (2):
  - Hospital Padre Hurtado, Santiago
  - Hospital Carlos Van Buren, Valparaíso
- Fundación Oftalmológica de Santander, Bucaramanga, Santander Department, Colombia
- Unidad Medica para la Salud Integral, San Nicolás de los Garza, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at sites in the United States, Brazil, Chile, Colombia, and Mexico, from 29 January 2021 (first participant enrolled to receive the study drug) to 28 January 2022 (last participant completed).
Pre-assignment Details: 78 participants with Coronavirus Disease 2019 (COVID-19) who were hospitalized were screened of which 57 were randomized in 1:1 ratio to receive either Alpha1-Proteinase Inhibitor (PI) (Human) plus Standard Medical Treatment (SMT) or placebo plus Standard Medical Treatment.
Groups:
- Alpha1-Proteinase Inhibitor + Standard Medical Treatment: Participants received the first intravenous (IV) infusion of liquid alpha1-proteinase inhibitor (human) 120 milligrams per kilogram (mg/kg), based on body weight on Day 1, followed by second liquid alpha1-proteinase inhibitor (human) dose of 120 mg/kg based on body weight, on Day 8 (second dose was not mandatory and was given at the principal investigator's [PI] discretion). Participants also received all standard of care interventions while hospitalized, from Day 1 to Day 29.
Period: Overall Study
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Started | 29 | 28
Safety Population (Safety population included all participants who received at least any amount of liquid Alpha1-PI (Human) plus SMT or placebo plus SMT.) | 27 | 27
Completed | 19 | 22
Not Completed | 10 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Death | 2 | 1
Not completed — Physician Decision (Does not Include Adverse Events) | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Reason Not Specified | 4 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all participants who were randomized.
Groups:
- Alpha1-Proteinase Inhibitor + Standard Medical Treatment: Participants received the first IV infusion of liquid alpha1-proteinase inhibitor (human) 120 mg/kg, based on body weight on Day 1, followed by second liquid alpha1-proteinase inhibitor (human) dose of 120 mg/kg based on body weight, on Day 8 (second dose was not mandatory and was given at the PI's discretion). Participants also received all standard of care interventions while hospitalized, from Day 1 to Day 29.
- Total: Total of all reporting groups
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (14.46) | 51.2 (12.14) | 51.7 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 15 | 17 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 10 | 24
  Not Hispanic or Latino | 15 | 18 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 22 | 21 | 43
  Race: Black or African American | 1 | 5 | 6
  Race: Asian | 3 | 0 | 3
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Dying or Requiring Intensive Care Unit (ICU) Admission
Time Frame: Up to Day 29
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 29 | 28
percentage of participants
  Percentage of Participants Dying | 6.9 | 3.6
  Percentage of Participants Requiring ICU Admission | 20.7 | 14.3
Statistical Analysis 1: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Percentage of Participants Dying; Test type: Superiority; Difference in percentages = 3.3
Statistical Analysis 2: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Percentage of Participants Requiring ICU Admission; Test type: Superiority; Difference in percentages = 6.4

2. Primary Outcome: Percentage of Participants Who Are Dependent on High Flow Oxygen Devices or Invasive Mechanical Ventilation
Time Frame: Day 29
Population: ITT population included all participants who were randomized. Percentage of participants are rounded off to the single decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 29 | 28
percentage of participants
  Dependent on High Flow Oxygen Devices | 6.9 | 0.0
  Dependent on Invasive Mechanical Ventilation | 3.4 | 0.0
Statistical Analysis 1: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Percentage of Participants Who are Dependent on High Flow Oxygen Devices; Test type: Superiority; Difference in percentages = 6.9
Statistical Analysis 2: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Percentage of Participants Who are Dependent on Invasive Mechanical Ventilation; Test type: Superiority; Difference in percentages = 3.4

3. Secondary Outcome: Change From Baseline in National Early Warning Score (NEWS)
Description: NEWS is clinical scoring developed to improve detection of deterioration in ill participant. It is based on 7 clinical parameters: Respiration rate, oxygen saturation, supplemental oxygen, systolic blood pressure (BP), pulse rate, level of consciousness, and temperature. A score of 0 and 2 was allocated to supplemental oxygen, 0 and 3 for level of consciousness and score of 0, 1, 2 and 3 for remaining parameters (i.e. respiration rate, oxygen saturation, systolic BP, pulse rate and temperature) where 0 = normal health condition to 3 = worst health condition; Higher scores indicated more severity. All scores were summed to get an aggregate score. Aggregate NEWS score ranged from 0 to 20, with higher scores indicating more severity/higher risk.
Time Frame: Baseline, Days 15 and 29
Population: ITT population included all participants who were randomized. Overall number analyzed are the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 18 | 22
score on a scale
  Change From Baseline at Day 15: number analyzed (Participants) | 18 | 21
  Change From Baseline at Day 15 | -1.1 (3.71) | -2.3 (2.22)
  Change From Baseline at Day 29: number analyzed (Participants) | 17 | 22
  Change From Baseline at Day 29 | -2.9 (2.38) | -2.5 (1.95)
Statistical Analysis 1: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Day 15; Test type: Superiority; p = 0.1453, Kenward-Roger — P-value was calculated using restricted maximum likelihood with the Kenward-Roger method for calculating the denominator degrees of freedom; Least Squares (LS) Mean Difference = 1.22, 95% CI 2-sided [-0.43 to 2.87]
Statistical Analysis 2: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Day 29; Test type: Superiority; p = 0.8015, Kenward-Roger — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 0.21, 95% CI 2-sided [-1.44 to 1.86]

4. Secondary Outcome: Time to Clinical Response as Assessed by NEWS Score ≤ 2 Maintained for 24 Hours
Description: Time to clinical response was reported at 50th percentile in days.
Time Frame: Up to Day 29
Population: ITT population included all participants who were randomized. Overall number analyzed are the participants who achieved clinical response.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 5 | 10
days | NA [NA to NA] — Median, upper and lower limit of 95% Confidence Interval (CI) was not estimable due to the number of participants with events much lower than 50%. | NA [5 to NA] — Median and upper limit of 95% CI was not estimable due to the number of participants with events lower than 50%.

5. Secondary Outcome: Time to Hospital Discharge
Description: Time to hospital discharge is defined as duration of hospitalization from Day 1 through Day 29.
Time Frame: Up to Day 29
Population: ITT population included all participants who were randomized. Overall number of participants analyzed signifies the number of participants with available data for analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 27 | 27
days | 5.0 [1 to 29] | 5.0 [2 to 29]
Statistical Analysis 1: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Test type: Superiority; p = 0.5135, ANOVA — P-value was calculated using an analysis of variance (ANOVA) model, including the length of hospital stay (days) as a dependent variable and treatment group as a fixed effect; LS Mean Difference of Duration = 1.48, 95% CI 2-sided [-3.04 to 6.00]

6. Secondary Outcome: Duration of ICU Stay
Description: Duration of ICU stay in days is analyzed for participants admitted to ICU post randomization.
Time Frame: Up to Day 29
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 27 | 27
days | 0.0 [0 to 29] | 0.0 [0 to 29]
Statistical Analysis 1: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Test type: Superiority; p = 0.1221, ANOVA — P-value was calculated using an ANOVA model, including the number of days in the ICU as a dependent variable and treatment group as a fixed effect; LS Mean Difference of Duration = 3.41, 95% CI 2-sided [-0.94 to 7.76]

7. Secondary Outcome: Duration of Any Oxygen Use
Time Frame: Up to Day 30
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 27 | 27
days | 7.0 [0 to 30] | 6.0 [0 to 30]
Statistical Analysis 1: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Test type: Superiority; p = 0.3329, ANOVA — P-value was calculated using an ANOVA model, including the number of days on oxygen as a dependent variable and treatment group as a fixed effect; LS Mean Difference of Duration = 2.78, 95% CI 2-sided [-2.92 to 8.48]

8. Secondary Outcome: Duration of Mechanical Ventilation
Description: Duration of Mechanical Ventilation is analyzed for participants requiring mechanical ventilation post randomization.
Time Frame: Up to Day 29
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 27 | 27
days | 0.0 [0 to 29] | 0.0 [0 to 28]
Statistical Analysis 1: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Test type: Superiority; p = 0.1092, ANOVA — P-value was calculated using an ANOVA model, including the number of days on mechanical ventilation as a dependent variable and treatment group as a fixed effect; LS Mean Difference of Duration = 3.48, 95% CI 2-sided [-0.81 to 7.77]

9. Secondary Outcome: Mean Change From Baseline in Ordinal Scale
Description: The ordinal scale is a 7-point scale ranging from 1 to 7 used to measure clinical status based on the following points: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities. Higher score indicated no severe illness. Mean change in Ordinal scale was evaluated by fitting a linear mixed-effects model for repeated measures (MMRM).
Time Frame: Baseline, Days 15 and 29
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 27 | 27
score on a scale
  Change From Baseline at Day 15 | 1.58 [1.00 to 2.15] | 2.21 [1.64 to 2.78]
  Change From Baseline at Day 29 | 1.80 [1.23 to 2.37] | 2.66 [2.09 to 3.22]
Statistical Analysis 1: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Day 15; Test type: Superiority; p = 0.1189, Kenward-Roger — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.63, 95% CI 2-sided [-1.43 to 0.17]
Statistical Analysis 2: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Day 29; Test type: Superiority; p = 0.0341, Kenward-Roger — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.85, 95% CI 2-sided [-1.64 to -0.07]

10. Secondary Outcome: Absolute Change From Baseline in Ordinal Scale
Description: The ordinal scale is a 7-point scale ranging from 1 to 7 used to measure clinical status based on the following points: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or ECMO; 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities. Higher score indicated no severe illness.
Time Frame: Baseline, Days 15 and 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 21 | 23
score on a scale
  Change From Baseline at Day 15: number analyzed (Participants) | 20 | 22
  Change From Baseline at Day 15 | 1.5 (1.96) | 2.3 (1.67)
  Change From Baseline at Day 29 | 1.8 (1.87) | 2.7 (1.48)

11. Secondary Outcome: Percentage of Participants in Each Severity Category of the 7-point Ordinal Scale
Description: The ordinal scale is a 7-point scale ranging from 1 to 7 used to measure clinical status based on the following points: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or ECMO 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities. The percentages are rounded off to the single decimal point.
Time Frame: Day 15 and Day 29
Population: ITT population included all participants who were randomized. Overall number of participants analyzed are unique number of participants with available data for analysis. Number analyzed are unique number of participants out of all the assessed participants with data available at the specified timepoint. Different participants may have contributed data for each timepoint. Participants who died during the study were assigned a value of 1 for the ordinal scale at every timepoint after the death.
Measure: Number; unit: percentage of participants
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 21 | 24
percentage of participants
  Day 15: Death: number analyzed (Participants) | 20 | 22
  Day 15: Death | 5.0 | 4.5
  Day 15: Hospitalized, on invasive mechanical ventilation or ECMO: number analyzed (Participants) | 20 | 22
  Day 15: Hospitalized, on invasive mechanical ventilation or ECMO | 10.0 | 0.0
  Day 15: Hospitalized, on non-invasive ventilation or high flow oxygen devices: number analyzed (Participants) | 20 | 22
  Day 15: Hospitalized, on non-invasive ventilation or high flow oxygen devices | 5.0 | 4.5
  Day 15: Hospitalized, requiring supplemental oxygen: number analyzed (Participants) | 20 | 22
  Day 15: Hospitalized, requiring supplemental oxygen | 10.0 | 4.5
  Day 15: Hospitalized, not requiring supplemental oxygen: number analyzed (Participants) | 20 | 22
  Day 15: Hospitalized, not requiring supplemental oxygen | 0.0 | 4.5
  Day 15: Not hospitalized, limitation on activities: number analyzed (Participants) | 20 | 22
  Day 15: Not hospitalized, limitation on activities | 25.0 | 22.7
  Day 15: Not hospitalized, no limitations on activities: number analyzed (Participants) | 20 | 22
  Day 15: Not hospitalized, no limitations on activities | 45.0 | 59.1
  Day 29: Death: number analyzed (Participants) | 21 | 23
  Day 29: Death | 9.5 | 4.3
  Day 29: Hospitalized, on invasive mechanical ventilation or ECMO: number analyzed (Participants) | 21 | 23
  Day 29: Hospitalized, on invasive mechanical ventilation or ECMO | 0.0 | 0.0
  Day 29: Hospitalized, on non-invasive ventilation or high flow oxygen devices: number analyzed (Participants) | 21 | 23
  Day 29: Hospitalized, on non-invasive ventilation or high flow oxygen devices | 4.8 | 0.0
  Day 29: Hospitalized, requiring supplemental oxygen: number analyzed (Participants) | 21 | 23
  Day 29: Hospitalized, requiring supplemental oxygen | 4.8 | 0.0
  Day 29: Hospitalized, not requiring supplemental oxygen: number analyzed (Participants) | 21 | 23
  Day 29: Hospitalized, not requiring supplemental oxygen | 0.0 | 0.0
  Day 29: Not hospitalized, limitation on activities: number analyzed (Participants) | 21 | 23
  Day 29: Not hospitalized, limitation on activities | 38.1 | 17.4
  Day 29: Not hospitalized, no limitations on activities: number analyzed (Participants) | 21 | 23
  Day 29: Not hospitalized, no limitations on activities | 42.9 | 78.3

12. Secondary Outcome: Time to Sustained Normalization of Temperature
Description: Time to sustained normalization of temperature was reported at 50th percentile in days.
Time Frame: Up to Day 29
Population: ITT population included all participants who were randomized. Participants who achieved sustained normalization of temperature were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 13 | 12
days | 7 [3 to NA] — Upper limit of 95% CI was not estimable due to insufficient participants with events. | NA [4 to NA] — Median and upper limit of 95% CI was not estimable due to the number of participants with events lower than 50%.

13. Secondary Outcome: Percentage of Participants Who Experienced Sustained Normalization of Fever
Description: Normalization of fever is defined as temperature < 36.6 °C armpit, < 37.2 °C oral, or < 37.8 °C rectal sustained for at least 24 hours.
Time Frame: Up to Day 29
Population: ITT population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 29 | 28
percentage of participants | 44.8 [26.4 to 64.3] | 42.9 [24.5 to 62.8]
Statistical Analysis 1: Comparison: Alpha1-Proteinase Inhibitor + Standard Medical Treatment vs Placebo + Standard Medical Treatment; Test type: Superiority; p = 0.8809, Chi-squared — P-value was calculated using Chi-square test with 5% level of significance to test the null hypothesis of no difference in the percentages of participants experiencing sustained normalization of fever; Difference in percentages = 1.9, 95% CI 2-sided [-24.1 to 28.3]

14. Secondary Outcome: Number of Participants Who Develop Acute Respiratory Distress Syndrome (ARDS)
Description: ARDS was defined based on Berlin criteria (chest imaging, origin of edema, oxygenation).
Time Frame: Up to Day 29
Population: ITT population included all participants who were randomized. Overall number of participants analyzed are the participants assessed for ARDS by Berlin criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 17 | 21
Participants | 5 | 2

15. Secondary Outcome: Time to Clinical Progression
Description: Time to clinical progression is defined as the time to death, mechanical ventilation, or ICU admission. Time to clinical progression was reported at 50th percentile in days.
Time Frame: Up to Day 29
Population: ITT population included all participants who were randomized. Overall number of participants analyzed are the participants with clinical progression.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alpha1-Proteinase Inhibitor + Standard Medical Treatment | Placebo + Standard Medical Treatment
Number analyzed (Participants) | 6 | 4
days | NA [NA to NA] — Median, Upper and Lower Limit of 95% CI was not estimable due to the number of participants with events much lower than 50%. | NA [NA to NA] — Median, Upper and Lower Limit of 95% CI was not estimable due to the number of participants with events much lower than 50%.

ADVERSE EVENTS:
Time Frame: Up to 90 days
Description: All-cause mortality: ITT population included all participants who were randomized.
  Adverse events: Safety population included all participants who received at least any amount of liquid Alpha1-PI (Human) plus SMT or placebo plus SMT.
Groups:
- Alpha1-Proteinase Inhibitor+Standard Medical Treatment: Participants received the first IV infusion of liquid alpha1-proteinase inhibitor (human) 120 mg/kg, based on body weight on Day 1, followed by second liquid alpha1-proteinase inhibitor (human) dose of 120 mg/kg based on body weight, on Day 8 (second dose was not mandatory and was given at the PI's discretion). Participants also received all standard of care interventions while hospitalized, from Day 1 to Day 29.
- Placebo+Standard Medical Treatment: Participants received IV infusions of 0.9% normal saline of commensurate volume to that of liquid alpha1-proteinase inhibitor as placebo on Day 1 and Day 8 (Day 8 was not mandatory and was given at the PI's discretion). Participants also received all standard of care interventions while hospitalized, from Day 1 to Day 29.
Arm/Group | Alpha1-Proteinase Inhibitor+Standard Medical Treatment | Placebo+Standard Medical Treatment
All-Cause Mortality (participants affected / at risk) | 2/29 | 1/28
Serious Adverse Events (participants affected / at risk) | 5/27 | 5/27
Other Adverse Events (participants affected / at risk) | 2/27 | 8/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha1-Proteinase Inhibitor+Standard Medical Treatment (N=27) | Placebo+Standard Medical Treatment (N=27)
Tracheal injury (Injury, poisoning and procedural complications) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha1-Proteinase Inhibitor+Standard Medical Treatment (N=27) | Placebo+Standard Medical Treatment (N=27)
Bradycardia (Cardiac disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Pneumonia bacterial (Infections and infestations) | 2 | 0
Blood pressure increased (Investigations) | 0 | 2

LIMITATIONS AND CAVEATS:
Study was early terminated due to lack of efficacy (futility).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT04547140/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT04547140/SAP_001.pdf